

#### **Informed Consent**

# INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH

A pilot study to evaluate the diagnostic performance of pleural touch preparations in pleuroscopy, a prospective study

| 2017-0746 | |
|-------------------------------|-----------------------|
| Study Chair: Horiana B. Grosu | |
| Participant's Name | Medical Record Number |

This is an informed consent and authorization form for a research study. It includes a summary about the study. A more detailed description of procedures and risks is provided after the summary.

## **STUDY SUMMARY**

The goal of this research study is to learn how accurately a type of lab testing called rapid on-site cytology examination (ROSE) can predict if pleural (lining of the lung) biopsy samples collected during an already-scheduled pleuroscopy will be malignant (cancerous).

ROSE testing is done by a specialist who will look at the biopsy samples during your procedure and determine if the sample is cancerous or not. This type of testing is a preliminary (early) result and has its own limitations. The ROSE testing results will be compared with final, lab results (which will be available in 2-3 business days) after the biopsy. Researchers want to learn if the ROSE testing results match the final lab results.

**This is an investigational study.** Pleuroscopy and ROSE testing are both FDA approved and commercially available. Both of these procedures will be done even if you do not take part in this study as part of your regular care. It is considered investigational to collect data about the results of the pleuroscopy and ROSE testing.

Future patients may benefit from what is learned. There are no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including potential expenses and time commitment.

You can read a list of potential side effects below in the Possible Risks section of this consent.

Your active participation in this study will be over after your tissue samples are collected and sent for testing.

You and/or your insurance provider will be responsible for the cost of the pleuroscopy and ROSE testing.

You may choose not to take part in this study. You may choose to have a pleuroscopy and ROSE testing without taking part in this study.

### 1. STUDY DETAILS

Up to 200 participants will take part in this multicenter study. Up to 100 be enrolled at MD Anderson.

# **Pleuroscopy**

If you agree to take part in this study, you will have a pleuroscopy to biopsy the lining of the lung as part of your standard care. You will receive a separate consent form describing the pleuroscopy and its risks.

After the biopsy sample is collected, the sample will be send to the pathology lab at MD Anderson for ROSE testing.

Depending on what your doctor thinks is in your best interest, you may not receive the ROSE results. However, you will receive the final lab results.

# **Medical Information**

Your medical information will be collected as part of this study. This information may include demographic information (such as your age and sex), information about your smoking history, your medical history, your current drugs, and/or laboratory test and imaging scan results.

This information will be collected from your medical record after the pleuroscopy procedure is performed. It will be stored in a password-protected computer server at MD Anderson.

#### 2. POSSIBLE RISKS

While on this study, you are at risk for side effects. You should discuss these with the study doctor. The known side effects are listed in this form, but they will vary from person to person.

There are no expected risks from the **ROSE testing of touch prep testing**.

Although every effort will be made to keep **study data** safe, there is a chance that your personal health information could be lost or stolen. All study data will be stored in password-protected computers and/or locked file cabinets. The study data will be stored in REDcap (a secure, web-based program used to collect data for research studies).

This study may involve unpredictable risks to the participants.

#### 3. COSTS AND COMPENSATION

If you suffer injury as a direct result of taking part in this study, MD Anderson health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. You will not be reimbursed for expenses or compensated financially by MD Anderson for this injury. You may also contact the Chair of MD Anderson's IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

Samples that are collected from you in this study may be used for the development of treatments, devices, new drugs, or patentable procedures that may result in commercial profit.

There are no plans to compensate you for any patents or discoveries that may result from your participation in this research.

You will receive no compensation for taking part in this study.

# **Additional Information**

4. You may ask the study chair (Dr. Horiana B. Grosu, at 713-792-6238) any questions you have about this study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB - a committee that reviews research studies) at 713-792-6477 with any questions that have to do with this study or your rights as a study participant.

- 5. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you decide you want to stop taking part in the study, it is recommended for your safety that you first talk to your doctor. If you withdraw from this study, you can still choose to be treated at MD Anderson.
- This study or your participation in it may be changed or stopped without your consent at any time by the study chair, the U.S. Food and Drug Administration (FDA), the Office for Human Research Protections (OHRP), or the IRB of MD Anderson.
- 7. You will be informed of any new findings or information that might affect your willingness to continue taking part in the study and you may be asked to sign another informed consent and authorization form stating your continued willingness to participate in this study.
- 8. MD Anderson may benefit from your participation and/or what is learned in this study.

# **Future Research**

#### Data

Your personal information is being collected as part of this study. These data may be used by researchers at MD Anderson and/or shared with other researchers and/or institutions for use in future research.

#### Samples

Samples (such as blood and/or tissue) are being collected from you as part of this study. Researchers at MD Anderson may use any leftover samples that are stored at MD Anderson in future research.

Before being used or shared for future research, every effort will be made to remove your identifying information from any data and/or research samples. If all identifying information is removed, you will not be asked for additional permission before future research is performed.

In some cases, all of your identifying information may not be removed before your data or research samples are used for future research. If future research is performed at MD Anderson, the researchers must get approval from the Institutional Review Board (IRB) of MD Anderson before your data and/or research samples can be used. At that time, the IRB will decide whether or not further permission from you is required. The IRB is a committee of doctors, researchers, and community members that is responsible for protecting study participants and making sure all research is safe and ethical.

If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data and/or samples.

#### Genetic Research

Research samples collected from you as part of this study may be used for genetic research, which may include whole genome sequencing. Whole genome sequencing is a type of testing in which researchers study your entire genetic makeup (DNA). This may help researchers learn how changes in the ordering of genes may affect a disease or response to treatment. If genetic research is done with your samples, those who have access to those samples may be able to identify you. The results of this research may also be able to be linked to you.

# **Authorization for Use and Disclosure of Protected Health Information (PHI):**

- A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
  - The IRB and officials of MD Anderson
  - Study monitors and auditors who verify the accuracy of the information
  - Individuals who put all the study information together in report form
- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible (according to state and federal law). However, in some situations, the FDA could be required to reveal the names of participants.
  - Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.
- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.
- E. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# **CONSENT/AUTHORIZATION**

I understand the information in this consent form. I have had a chance to read the

| consent form for this study, or have had it read to me. I have had about it, ask questions, and talk about it with others as needed. I permission to enroll me on this study. By signing this consent for any of my legal rights. I will be given a signed copy of this conser | give the study chair<br>m, I am not giving up |
|---|---|
| SIGNATURE OF PARTICIPANT | DATE |
| PRINTED NAME OF PARTICIPANT | |
| LEGALLY AUTHORIZED REPRESENTATIVE (LAR) The following signature line should only be filled out when the pathe capacity to legally consent to take part in the study and/or signature or her own behalf. | • |
| SIGNATURE OF LAR | DATE |
| PRINTED NAME and RELATIONSHIP TO PARTICIPANT | _ |
| WITNESS TO CONSENT I was present during the explanation of the research to be perform 2017-0746. | ned under Protocol |
| SIGNATURE OF WITNESS TO THE VERBAL CONSENT PRESENTATION (OTHER THAN PHYSICIAN OR STUDY CHAIR A witness signature is only required for vulnerable adult participants. If witness participant, leave this line blank and sign on the witness to assent page instead | ing the assent of a pediatric |
| PRINTED NAME OF WITNESS TO THE VERBAL CONSENT | _ |
| PERSON OBTAINING CONSENT I have discussed this research study with the participant and/or his representative, using language that is understandable and appropriate fully informed this participant of the nature of this study and and risks and that the participant understood this explanation. | oriate. I believe that I |
| PERSON OBTAINING CONSENT | DATE |
| PRINTED NAME OF PERSON OBTAINING CONSENT | |

| TRANSLATOR TRANSLATOR |
|---|
| have translated the above informed consent as written (without additions or subtractions) intoand assisted the people |
| (Name of Language) obtaining and providing consent by translating all questions and responses during the |
| consent process for this participant. |
| NAME OF TRANSLATOR SIGNATURE OF TRANSLATOR DATE |
| ☐ Please check here if the translator was a member of the research team. (If checked, a witness, other than the translator, must sign the witness line below.) |
| SIGNATURE OF WITNESS TO THE VERBAL TRANSLATION DATE (OTHER THAN TRANSLATOR, PARENT/GUARDIAN, OR STUDY CHAIR) |

PRINTED NAME OF WITNESS TO THE VERBAL TRANSLATION